CLINICAL TRIAL: NCT04791865
Title: Pediatric HIV Disclosure Benefits Study (PhD-BS) - Sankofa 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H-44300; 1R01HD103512-01 (NIH)
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: HIV
Keywords: resources limited settings; HIV infected children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): During the control period, patients and caregivers recruited at the clinics will receive the current practice in the clinic, where the health care provider is expected to assess the caregiver and child readiness for disclosure during clinic appointments and give some information as they think indicated.
  Interventions: Behavioral: Usual Care
- Disclosure intervention (Experimental): Participants who are assigned to the Sankofa intervention will take part in the process of disclosure (pre-disclosure, disclosure, and post-disclosure phases) with the adherence and disclosure specialist (ADDS).
  Interventions: Behavioral: Disclosure intervention

INTERVENTIONS:
Behavioral: Disclosure intervention — Participants who are assigned to the Sankofa intervention will take part in the process of disclosure (pre-disclosure, disclosure, and post-disclosure phases) with the adherence and disclosure specialist (ADDS).
  Arms: Disclosure intervention
Behavioral: Usual Care — During the control period, patients and caregivers recruited at the clinics will receive the current practice in the clinic, where the health care provider is expected to assess the caregiver and child readiness for disclosure during clinic appointments and give some information as they think indicated.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to conduct a pragmatic, stepped wedge cluster randomized trial in 12 HIV pediatric clinics in Ghana to determine effectiveness, health benefits, cost and implementation to inform scale-up and sustainability of pediatric disclosure.

DETAILED DESCRIPTION:
In this 5-year study, the investigators would like to build upon the successful Sankofa trial by testing the intervention in a larger scale study delivered in "real-world" clinic conditions over time in Ghana.

The purpose of this study is to conduct a pragmatic, stepped wedge cluster randomized trial in 12 HIV pediatric clinics in Ghana to determine effectiveness, health benefits, cost and implementation to inform scale-up and sustainability of pediatric disclosure. The study will recruit dyads of 720 children (ages 7-18) and their caregivers from twelve (12) clinics, which will be randomly assigned to each of the four roll-out schedules ("wedge steps"), with three clinics per step.

The two groups in the study are usual care and disclosure intervention. During the control period, patients and caregivers recruited at the clinics will receive the current practice in the clinic, where the health care provider is expected to assess the caregiver and child readiness for disclosure during clinic appointments and give some information as they think indicated. No formal pediatric disclosure guidelines or educational materials exist in Ghana.

During the intervention period, the manualized, with standard operation procedures, Sankofa intervention will be delivered. The intervention is guided by the disclosure model and contains key elements to target well-documented, modifiable barriers to promote disclosure.

The primary outcome is disclosure after one year (48 weeks) of the intervention. Secondary outcomes are antiretroviral medication adherence, health (virologic, immunologic, psychosocial, behavioral), cost, and implementation.

The trial will be conducted with a strong team of interdisciplinary investigators at two universities in Ghana, Yale and Johns Hopkins University in partnership with the Ghana Ministry of Health (MoH), Ghana Health Service (GHS) and a community advisory board.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected children
* Children between the ages of 7-18 who do not know their HIV diagnosis (based on caregiver account and medical records confirmation) and their caregivers will be eligible to participate in the study

Exclusion Criteria:

* HIV-infected children less than 7 years
* HIV-infected children with congenital or developmental disorders
* HIV-infected children with comorbidities such as sickle cell disease or diabetes that require frequent clinic visits or hospitalizations
* Children with AIDS-defining illness or end stage AIDS.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 747 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
HIV disclosure rate | 1 year after intervention
  Structured and caregiver-centered and culturally-relevant disclosure intervention will be delivered by an adherence and disclosure specialist to the caregiver. After one year, the rate of disclosure of the HIV status of the children will be assessed.

SECONDARY OUTCOMES:
Change in Antiretroviral medication adherence | 5 year
  Medication adherence will be assessed with the AIDS Clinical Trials Group (ACTG) Adherence Questionnaire self-report questionnaire. This will be assessed every 3 months up until end of study. This measures provides a ratio of adherence to antiviral medication requirements. A score of 1 equals perfect adherence and 0 represents no adherence.
Antiretroviral medication adherence - Pharmacy refill measurement | 5 year
  The pharmacy-based time-to-refill measure adherence is calculated as the number of months for which antiretroviral therapy claims were submitted to the pharmacy, divided by the number of complete months during the period under consideration, and the results multiplied by 100
Antiretroviral medication adherence - HIV-1 RNA | 5 year
  HIV-1 RNA is calculated by
Immunologic health | 5 year
  The immunologic staging of their disease according to both the U.S. CDC and WHO classification criteria will be used to determine immunologic health using patient's medical chart.
Behavioral health - CBCL child version | 5 year
  Children health will be measured by using the Child Behavior checklist-child version (CBCL). For each item on the CBCL, the respondent is asked to choose from a three-point response scale indicating whether a problem behavioral description is "not true" (= 0), "somewhat or sometimes true" (= 1), or "very true or often true" (= 2) of the child
Behavioral health - CBCL parent version | 5 year
  Children health will be measured by using the Child Behavior checklist-child version (CBCL). For each item on the CBCL, the respondent is asked to choose from a three-point response scale indicating whether a problem behavioral description is "not true" (= 0), "somewhat or sometimes true" (= 1), or "very true or often true" (= 2) of the child
Child Depression Inventory (CDI) | 5 year
  The CDI is an 27 item questionnaire on a three-point scale to assess depression symptoms. The cumulative score will be calculated
Beck Depression Inventory | 5 year
  The Caregiver's psychosocial health will be measured with the 21-item Beck Depression Inventory (BDI). The Beck Depression Inventory (BDI) is a 21-item, multiple-choice inventory. Respondents are asked to rate each item based on four response choices according to the severity of the symptoms, ranging from the absence of a symptom to an intense level, during the past week. BDI scores from 0 through 9 indicate no or minimal depression; scores from 10 through 18 indicate mild to moderate depression; scores from 19 through 29 indicate moderate to severe depression; and scores from 30 through 63 indicate severe depression.
Implementation - Retention | 5 year
  Proportion of subjects retained throughout the implementation phase. This will be reported >90%, 60-90%, and <60%)
Implementation - Caregiver 6-month log | 6 month
  The caregivers' 6-month surveys (e.g., caregivers' experience summarized into 3 categories: 1=Not Satisfactory, 2=Satisfactory, 3=Very Satisfactory). will be used to characterize a composite outcome for implementation success: 1= successful, 2= intermediate, 3= problematic
Incremental cost-effectiveness ratio | 5 year
  The incremental cost effectiveness ratio (ICER) will be used to compare pediatric intervention relative to the standard of care to assess cost-effectiveness. The 1 year ratio will provide directly observed near term economic impact of disclosure.
Change in HIV -1 RNA Viral Load | 5 years
  The HIV-1 RNA viral load will be measured every 6 months to determine the change over 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Paintsil, MD, FAAP, Principal Investigator — Boston University Chobanian & Avedisian School of Medicine, Pediatrics; Veronika Shabanova, PhD, Principal Investigator — Yale University, Pediatrics, Biostatistician
Locations (1):
- Korle-Bu Teaching Hospital, Accra, Ghana

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Afrane AKA, Bobbala A, Martyn-Dickens C, Renner L, Antwi S, Kusah JT, Amissah K, Quaye D, Bosomtwe D, Gan G, Parziale S, Reynolds NR, Paintsil E, Shabanova V; Sankofa Study Team. Changes in caregiver psychosocial factors known to affect pediatric HIV disclosure: the Sankofa clinical trial experience in Ghana (2013-2023). AIDS Care. 2025 Dec 2:1-16. doi: 10.1080/09540121.2025.2594607. Online ahead of print. PMID 41330401
- [Derived] Reynolds NR, Shabanova V, Renner L, Antwi S, Ayisi Addo S, Enimil AK, Lartey M, Gan G, Parziale S, Aikins Amissah K, Kusah JT, Ofori-Atta AL, Slade E, Agyarko-Poku T, Paintsil E. Scale-up of a paediatric HIV disclosure intervention in Ghana using a stepped wedge cluster randomised trial design: Sankofa 2 protocol and implementation. BMJ Open. 2025 Nov 13;15(11):e099681. doi: 10.1136/bmjopen-2025-099681. PMID 41238360